CLINICAL TRIAL: NCT01946464
Title: Novel Technique for Face Mask Ventilation
Status: Terminated | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: 2012001161
Record Dates: First submitted 2013-01-25; First posted 2013-09-19 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-07

CONDITIONS: Obstructive Sleep Apnea
Keywords: edentulous; bearded; patients; requiring; general anesthesia; Mallampati Class II or IV
MeSH Terms: conditions — Sleep Apnea, Obstructive; Mouth, Edentulous

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- undergoing surgery with general anesthesia: pts: edentulous, bearded, obstructive sleep apnea, Mallampati Class III or IV
- Mallampati I and II: Control group Mallampati I visualization of tonsils, uvula and soft palate Mallampati II visualization of hard and soft palate, and upper portion of tonsils and uvula.

SUMMARY:
This study is being done to see if we can improve the way we manage patients' airways. In some instances patients who have a beard, who do not have teeth or have breathing problems during sleep present a challenge to the anesthesiologist. In such patients, it is sometimes difficult to provide air/oxygen for breathing using a mask. The study doctors would like to investigate a new method for holding a mask on the face of those patients. They are interested in comparing a new method against two older methods. They believe the new method will deliver a larger amount of air to the lungs. This information may help doctors provide better care for patients who have beards, no teeth, or breathing problems during sleep.

DETAILED DESCRIPTION:
Goal: To demonstrate that a modified submandibular hand position can overcome shortcomings to the traditional E-C mask grip during difficult bag mask ventilation by a single practitioner.

Introduction:

Mask Ventilation is a vital skill that needs to be mastered by virtually all medical personnel. Whether in an acute care setting or a remote field situation, caregivers well trained in mask ventilation have the capacity to save lives. Therefore, any advances in this technique will have widespread and profound impact on morbidity and mortality outcomes.

Traditionally there are two main styles of mask ventilation, one-handed and two handed mask grips. After the initiation of one-handed mask ventilation, if the provider experiences difficulty, a switch is made to a two-handed grip. The two-handed grip has the disadvantage of requiring a second caregiver to provide tidal volumes to the patient in distress.

The traditional one-handed grip is taught using the "E" and "C" method. The most usual reason for failure to ventilate with this method is air leak on the side opposite the stabilizing hand.

The two-handed grip allows both hands to stabilize most of the circumference of the facemask. This is valuable because it can overcome an inadequate seal that is due to an unstable single-handed grip. Failure to obtain adequate seal between the face and a pliable facemask can also be attributed to variables not related to ventilation technique. For example, improper fit, patient anatomical variability, edentulousness, and full beard may also contribute to inadequate seal and deficient masked ventilation.

Han et al. have delineated the classification of a difficult airway using a four-point system, where grade 3 indicates difficult mechanical ventilation (inadequate, unstable, or requiring two providers) and grade 4 indicates impossible ventilation. Kheterpal et al. later showed that body mass index of 30 kg/m2 or greater, a beard, Mallampati classification III or IV, age of 57 yr or older, severely limited jaw protrusion, and snoring were independent risk factors for a grade 3 airway. Snoring and thyromental distance of less than 6 cm were shown to be independent risk factors for a grade 4 airway. Both studies utilized the traditional one-handed grip or a two-handed grip when attempting mechanical ventilation.

Given that some of the established risk factors in a difficult airway may be related to inadequate seal, it is crucial to explore limitations in the traditional methods of mask ventilation. For example, the traditional "C" and "E" one-handed grip only allows for the provider to apply pressure to the left border of the facemask. This leaves the right border of the facemask vulnerable to losing a seal and air escaping.

Here we propose a novel Sub Mandibular one-handed grip that allows for pressure to be applied to both the left and right borders of the facemask during masked ventilation. The anesthesia provider (AP) will stand perpendicular to the long axis of the patient's body, aligning the AP's umbilicus to the patient's mentum. Next, the AP will place their fifth digit along the body of the left mandible. The fourth digit will be placed along the body of the right mandible. The AP will rotate clockwise at the hip while keeping their elbow against their body to lift the patient's chin to 45 degrees. This rotational force adds strength to the chin lift maneuver. The AP will avoid pressing the soft tissue in the submental triangle. The first digit will be used to apply pressure to the left border of the facemask while the second and third digits will be used to apply pressure to the right border of the facemask. Accordingly, the provider will be able to apply pressure to both the left and right borders of the facemask with the intention of eliminating the right-sided air leak often observed while utilizing the traditional "C" and "E" one-handed technique.

A demonstration of each of the 3 grips will be shown to the qualifying AP either on an awake patient or a staff member. The AP will be asked to provide return demonstrations.

. After informed consent is obtained baseline vital signs will be documented. An intravenous line will be started and the American Society of Anesthesiologists (ASA) standard monitoring devices will be placed. Study subjects (n=6 in each) will be stratified into the following patient groups: edentulous, bearded, obstructive sleep apnea, Mallampati Class III or IV, and previous neck radiation.

Subjects assigned a Mallampati Class I or II with no comorbidities will serve as the control group (n=6). Mallampati Class I patients will be defined as those patients with clear visualization of the tonsils, uvula, and soft palate during inspection of the oral cavity by the provider. Mallampati Class II patients will be defined by visualization of the hard and soft palate, and upper portion of the tonsils and uvula. Mallampati Class III patients will be defined by visualization of the soft and hard palate, and base of the uvula. Mallampati Class IV patients will be defined by visualization of the hard palate only.

Two groups of anesthesia care providers, faculty and Advanced Practice Nurse Anesthesia (APN-A) (formerly known as Certified Registered Nurse Anesthetists/(CRNAs), will be asked to participate in the study. Data collected about the professional participants will include gender, dominant hand, grip strength and age range. These participants will be asked to use the hand dynamometer and their score will be recorded.

All patients will be undergoing standard IV induction of general anesthesia by anesthesiology attending staff with 2 μg/kg fentanyl and 2 mg/kg propofol, as well as 1 to 2mg of midazolam and 1mg/kg of lidocaine at the anesthesiologist's discretion. After loss of consciousness patients will receive 2 mg/kg of succinylcholine in preparation for intubation.

After induction of general anesthesia and before placement of the endotracheal tube (ETT) or laryngeal mask airway (LMA), the experienced anesthesia provider will attempt to ventilate the patient using an adult sized facemask. Each facemask will be pre-inflated with 150cc of room air and facemask will be placed over patient's oral cavity utilizing the traditional one-handed C and E technique. The anesthesia provider will then provide a chin lift maneuver to 45 degrees and activate the ventilator 45 seconds after succinylcholine administration. A preset tidal volume of 8cc/kg will be delivered for 8 breaths. Any air leak will be noted and provider will attempt to minimize air leak. Tidal volumes (TV), peak airway pressures(PAP) will be recorded at each breath by an independent observer as well as heart rate (HR), oxygen saturation rate (spO2) and presence/absence of Carbon dioxide ( + /- CO2).

The same process delivering 8 breaths with the same data parameter collection will be repeated using the novel sub mandibular grip followed by the two-handed grip. Each of the facemask techniques is estimated to take 1.5 minutes for a total 5 of minutes.

In the cases where tidal volume achieved is a level below 1cc/kg, an oral airway will be used, the ventilation reinstituted, and the provider will record a new set of data using the three techniques as described.

Rescue:

If the patient cannot be ventilated after placement of the oral airway, an endotracheal tube (ETT) will be placed following standard hospital protocol and the study for this patient will be terminated.

All providers will have experience of 12 months or greater in airway management. We will recruit anesthesia providers of both genders. Because grip strength can vary between providers we will measure grip strength using a dynamometer (BASELINE® Hydraulic Hand Dynamometer). The anesthesia providers' age range, gender, grip strength and hand size (tip of 2nd digit to wrist length) will be recorded. The AP will be tested with the dynamometer in the dominant hand. The arm will be held at the side of the body. The base of the dynamometers should rest at the heel of the palm while the handle should rest on the four fingers. The (AP) should squeeze the handle with maximum isometric effort, which is maintained for about 5 seconds. No other body movement is allowed. The AP will be encouraged to give a maximum effort. The AP grip strength in pounds will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* undergoing general anesthesia
* no longer have your own teeth
* have a beard
* have obstructive sleep apnea
* ASA score of 1, 2,3
* BMI<45
* Mallampati I, II. II or IV -(nil per os) Nothing taken orally for 8 hours-

Exclusion Criteria:

* ASA 4
* Morbidly obese >45
* Loose teeth
* cervical neck instability
* history of difficult airway
* Pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pts coming to Same Day Surgery who require anesthesia
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
tidal volume | at induction
  The primary aim of this study is to determine if using the novel one hand approach provides better ventilation as demonstrated by the tidal volumes.

SECONDARY OUTCOMES:
ventilation technique | at induction
  The secondary aim is to analyze the anesthesia providers' ability to ventilate using all three techniques based on their individual gender, grip strength, hand size and age range

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Grech, MD, Principal Investigator — Rutgers/NJMS
Locations (1):
- Rutgers RBHS Newark -DOC, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No